CLINICAL TRIAL: NCT00916981
Title: Treatment of Refractory Non-union Fractures by Pre-osteoblast Cells Grafting : a Pilot Study.
Brief Title: Treatment of Atrophic Nonunion by Preosteoblast Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jean-Philippe Hauzeur (Other)
Responsible Party: Sponsor-Investigator, Jean-Philippe Hauzeur, Principal investigator, University of Liege
Organization: University of Liege (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ref:2006-73
Record Dates: First submitted 2009-06-03; First posted 2009-06-10 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Pseudarthrosis; Fractures, Ununited
Keywords: pseudarthrosis; Treatment; osteoblast grafting; cell therapy; nonunion
MeSH Terms: conditions — Pseudarthrosis; Fractures, Ununited

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: percutaneous autologous preosteoblast cells implantation — percutaneously injection of preosteoblast into the nonunion under radioscopic control
  Other Names: PREOB

SUMMARY:
Treatment of nonunion, delayed union and malunion fractures of long bones remains problematic. The definition of nonunion is a failure of the fracture to heal in six months in a patient in whom progressive repair had not been observed radiographically between the third and sixth month after the fracture. First of all good surgical techniques are stable immobilization must be obtained and local sepsis excluded. Then stimulation of the callus is required. Numerous techniques have been developed ranging from invasive interventions (including internal fixation with the use of bone graft or bone graft substitutes) to non invasive procedures (ultrasound and pulsed electromagnetic fields).

Recently, autologous cell therapy was presented as an interesting approach. The concept of such therapies is based on the effect of stem cells presented in the bone marrow and able to be transformed in osteoblast cells. The percutaneous technique of autologous bone-marrow grafting is a minimally invasive alternative able to produce a good healing of the fracture. The efficacy is dependent of the concentration in progenitor cell reinjected. An optimization of this type of treatment could be achieved using a technique to increase the differentiation of the bone marrow cells in preosteoblasts before the injection in situ by an adequate culture. Therefore we would like to start a pilot open study on the feasibility and the efficacy of implantation of preosteoblasts into nonunion. Two different presentations exist: the atrophic and the hypertrophic pseudarthrosis in relationship with radiological features of bone proliferation at the tip of bone fragments. Some data support that atrophic and hypertrophic nonunion fractures could have different physiopathological factors. So, in a first time we only would evaluate the atrophic form and to determine in an open study the effect of the implantation of preosteoblasts into atrophic nonunion.

DETAILED DESCRIPTION:
We will recruit 30 patients having a atrophic nonunion fracture of long bone present for minimum 6 months.50 ml of bone marrow harvest will be performed under local anaesthesia 3 weeks before the implantation. After three weeks of culture, preosteoblastic cells will be injected into the site of pseudarthrosis under radioscopic control, using percutaneously a 3 mm trephine.

An immobilization and non weight-bearing of the bone will be respected during the first month after the injection. If callus could be observed on radiographs, partial mobilization and weight-bearing will be allowed during the second month.

ELIGIBILITY:
Inclusion Criteria:

* Fracture of a long bone having insufficient healing after minimum 6 months.
* Be able and willing to participate in the study.

Exclusion Criteria:

* Evidence of malignant disorder in the past five year.
* Patient who is positive for an HIV, hepatitis B or C infection.
* Insufficient reduction of the fracture with displaced fragments.
* Evidence of local sepsis by biological parameters and/or positive isotopic scan using leucocytes labelled by Indium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
radiological progression of bone fusion | 1, 2, 3, 4, 5, 6 months
  monthly

SECONDARY OUTCOMES:
reduction of pain using VAS | each month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Hauzeur, MD, PhD, Principal Investigator — University of Liège, Belgium
Locations (1):
- CHU Sart Tilman, Liège, Liège, Belgium